CLINICAL TRIAL: NCT02244138
Title: Improving Adolescent Health Outcomes Through Preventive Care Transformation
Acronym: AdolCHICA
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew Aalsma, Associate Professor, Indiana University
Other Study IDs: 1308038999; R01HS022681 (AHRQ)
Record Dates: First submitted 2014-09-12; First posted 2014-09-18 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Sexually Transmitted Diseases; Depression Diagnosis; Substance Use Disorders
Keywords: Adolescent; Screening; Primary Care; Computer Decision Support Systems
MeSH Terms: conditions — Sexually Transmitted Diseases; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescent CDSS: Implementation clinic site for CDDS
  Interventions: Behavioral: Adolescent CDSS

INTERVENTIONS:
Behavioral: Adolescent CDSS — computer decision support system (CDSS) for health care providers of adolescents in primary care

SUMMARY:
Preventive care for adolescents is vitally important for maximizing their health and well-being. Unfortunately, pediatric primary care frequently fails to meet the preventive needs of adolescents as demonstrated by poor health outcomes for this population.

In this grant application, the investigators propose to expand an existing computer decision support system (CDSS) into the investigators adolescent primary care practices for the purpose of implementing a comprehensive, and developmentally appropriate, screening and physician decision support process. Prior work completed by the investigators research group has demonstrated the feasibility of using CDSS to implement and evaluate clinical guidelines. The investigators seek to positively impact the effectiveness of preventative primary care visits by applying this previous success to the investigators adolescent practice. The investigators hypothesize that the implementation of developmentally appropriate universal screening practices, using tablet technology, and enhanced physician decision support regarding clinically relevant guidelines for all annual adolescent preventive care visits will result in better health outcomes, including higher rates of adherence to physician recommendations and improved patient functioning.

The specific research aims of this proposal are:

Aim 1: Expand and modify an existing CDSS to include an Adolescent Preventive Care Module comprised of developmentally appropriate screening tools for adolescents aged 11 to 21 years and tailored evidence-based clinical decision support for physicians.

Aim 2: Evaluate the impact of the Adolescent Preventive Care Module on the identification of specific mental and physical health problems and treatment outcomes in an adolescent primary health care setting.

Adolescent primary care issues of interest for this project include sexually transmitted infection (STI), depression, substance use and Human Papillomavirus (HPV) immunization. The investigators expect this project to improve the health outcomes of adolescents, guide future efforts to implement universal screening and CDSS in a variety of primary care settings, and provide additional evidence to support broad-based electronic screening and computerized decision support for use in preventive care as a method for improving adolescent health.

ELIGIBILITY:
Inclusion Criteria:

* 11-21 years
* attending primary care clinic

Exclusion Criteria:

* none

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent from primary care clinics will be studied
Sampling Method: Non-Probability Sample
Enrollment: 2831 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
sexually transmitted infection | 12 months
  diagnosis of sexually transmitted infection by physician as indicated in electronic health record for patient

SECONDARY OUTCOMES:
depression | 12 months
  diagnosis of depression by physician as indicated in electronic health record for patient

OTHER OUTCOMES:
substance use | 12 months
  diagnosis of substance use by physician as indicated in electronic health record for patient

CONTACTS AND LOCATIONS:
Overall Officials: matthew c aalsma, phd, Principal Investigator — Indiana University
Locations (1):
- Eskenazi Medical Group, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Aalsma M, Keys J, Ferrin S, Shan M, Garbuz T, Scott T, Adams Z, Hulvershorn L, Downs S. Adolescent suicide assessment and management in primary care. BMC Pediatr. 2022 Jul 2;22(1):389. doi: 10.1186/s12887-022-03454-4. PMID 35780090
- [Derived] Etter DJ, McCord A, Ouyang F, Gilbert AL, Williams RL, Hall JA, Tu W, Downs SM, Aalsma MC. Suicide Screening in Primary Care: Use of an Electronic Screener to Assess Suicidality and Improve Provider Follow-Up for Adolescents. J Adolesc Health. 2018 Feb;62(2):191-197. doi: 10.1016/j.jadohealth.2017.08.026. Epub 2017 Nov 28. PMID 29195764
- [Derived] Aalsma MC, Zerr AM, Etter DJ, Ouyang F, Gilbert AL, Williams RL, Hall JA, Downs SM. Physician Intervention to Positive Depression Screens Among Adolescents in Primary Care. J Adolesc Health. 2018 Feb;62(2):212-218. doi: 10.1016/j.jadohealth.2017.08.023. Epub 2017 Nov 23. PMID 29174939